CLINICAL TRIAL: NCT06360159
Title: Effect of Massage on Stress, Comfort and Health Parameters of Newborns Receiving Nasal CPAP
Brief Title: Massage for Newborns Receiving Nasal CPAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Besiktas (Other)
Responsible Party: Sponsor-Investigator, Sultan Besiktas, Principal Investigator, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Massage on Newborns
Record Dates: First submitted 2024-02-15; First posted 2024-04-11 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Massage; Stress; Newborn; Comfort
Keywords: massage; Stress; comfort; salivary cortisol level; nasal CPAP
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Intervention group (Massage): Babies in the intervention group will be massaged three times a day for 3 days, each session lasting 15 minutes, in accordance with the field massage technique. Massage application will be applied 1 hour after the babies are fed. For massage application, apply oil, solution and cream etc. to the baby's skin will not be used. During the massage application, the baby will be placed in prone and supine positions. Massage will be applied to the newborns in the intervention group by the assistant researcher.
  Control group: Apart from clinical routine practices, salivary cortisol samples will be taken from newborn babies in the control group and abdominal circumference of the babies will be measured.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): INTERVENTION GROUP: For newborn babies in the massage group; Field massage protocol will be used and the massage will be applied by the assistant researcher. Field massage developed by Field et al. (1986); In a standardized 15-minute stimulation session, the stimulation technique is changed every 5 minutes, and it is applied 3 times a day as tactile stimulation in the first 5 minutes, kinesthetic stimulation in the second 5 minutes and tactile stimulation in the third 5 minutes.(tactile stimulation-kinesthetic stimulation-tactile stimulation)
  Interventions: Other: Intervention
- Control Group (No Intervention): CONTROL GROUP: Apart from clinical routine practices, salivary cortisol samples will be taken from newborn babies in the control group and abdominal circumference of the babies will be measured.

INTERVENTIONS:
Other: Intervention — As an intervention, the newborn will be massaged.
  Arms: Intervention Group

SUMMARY:
One of the most frequently required treatments for respiratory distress in neonatal intensive care is continuous positive airway pressure (NCPAP) support through the nose. NCPAP application has many advantages but also disadvantages and complications.

Gastric-abdominal distension, which is a complication of NCPAP application, is caused by gas entering the stomach and gastrointestinal tract. Feeding intolerance may develop in the newborn due to abdominal distension. In recent studies, it has been determined that non-pharmacological methods and supportive developmental care practices used to increase the comfort and reduce pain and stress of babies who experience painful procedures such as NCPAP application and who are exposed to the stressful neonatal intensive care unit environment are effective in increasing comfort and reducing pain and stress. These practices include therapeutic touch, mother's voice, fetal position, white noise, lullaby, wrapping and massage. In the literature, a quasi-experimental study examining the effect of massage (Field massage technique) on the respiration, heart rate and oxygen saturation of 28-34 week old newborns with respiratory distress syndrome who received nasal CPAP showed that massage had no significant effect on oxygen saturation, but respiration and heart rate decreased after the massage. has been determined. There are studies in the literature examining the effects of therapeutic touch, mother's voice, fetal position, white noise, lullaby and wrapping in order to increase the comfort of newborns receiving nasal CPAP, reduce stress and pain, and prolong sleep time. However, no research has been found in the literature examining the effects of massage on the stress, comfort and health parameters of newborns receiving nasal CPAP.

DETAILED DESCRIPTION:
Purpose of the research

This research was planned to determine the effect of massage on stress (behavioral-newborn stress scale and biological-salivary cortisol level), comfort (Newborn Comfort Behavior Scale) and health parameters (bilirubin level, amount of food intake, abdominal distension and defecation frequency) of newborns receiving nasal CPAP. .

Research Type: This research is a randomized controlled experimental study.

Population and sample/Study group

The population of the research will consist of newborn babies admitted to the Neonatal Intensive Care Unit of Erzincan Binali Yıldırım University Mengücek Gazi Training and Research Hospital. The research sample will consist of newborns who meet the research inclusion criteria. In the literature review, no study was found that evaluated the effect of massage on babies' stress (behavioral-newborn stress scale, biological-salivary cortisol level), comfort and health parameters (bilirubin level, food intake amount, abdominal distension and defecation frequency). Asmarani et al. (2020) in their study examining the effect of massage on salivary cortisol levels in premature newborns, it was determined that they reached 39 (19 intervention group, 20 control group) newborns (Asmarani et al., 2020). In this study, it was decided that the number of newborns in the groups would be 18, based on α = 95% confidence level and 80% power. The research sample will consist of 36 newborns (18 intervention group, 18 control group) who meet the research inclusion criteria.

Data collection tools

Newborn Information Form: Diagnosis of the newborn baby, gender, type of birth, height, birth weight, gestational and postnatal age, Apgar score, day of admission and discharge, time to start nasal CPAP application, total time of receiving nasal CPAP application, the status of receiving phototherapy treatment and the total number of hours of phototherapy treatment during the study will be recorded on this form.

Follow-up Form: The newborn baby's 3-day bilirubin level, defecation frequency, food intake amount, salivary cortisol level, abdominal circumference, stress and comfort scores will be recorded in this form during the study period.

Phototherapy Device: Okuman (Bilicare-BC 050 000) brand phototherapy device with blue LED technology will be used for phototherapy.

Digital Electronic Scale: NECK brand EBSH model baby scale (20 kg capacity - 5 g precision) will be used to measure the body weight of newborn babies.

Camera: A camera that can record, has high resolution, and has high optical focus will be used to evaluate the stress and comfort levels of babies in the intervention and control groups. The flash feature of the camera will not be used so that the baby is not disturbed by the camera light.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age greater than 34 weeks
2. Birth weight of 2000 g and above,
3. Within the first 24 hours of nasal CPAP application
4. Fed at least one hour before the procedure,
5. Having no congenital anomaly,
6. Not having any disease at birth such as neonatal asphyxia, hemolytic condition, patent ductus arteriosus (PDA),
7. Those who have not undergone a surgical operation,
8. The mother does not have alcohol, cigarette or other drug addiction,
9. These are newborns to whom one of the parents (mother or father) has given verbal and written consent.

Exclusion Criteria:

1. Rh and ABO incompatibility,
2. APGAR score below 6,
3. Analgesic or anesthetic medication is administered for sedation,
4. Saliva sample cannot be taken,
5. NEC developing,
6. Leaving the hospital before the end of the working period,
7. Having had maternal obstetric complications,
8. Receiving blood transfusion during the study,
9. Newborns whose parents wish to withdraw from the study will not be accepted.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Stress Level | Every day of the study for 3 days, the newborn's stress level will be evaluated 5 minutes before the first massage application and 5 minutes after the third massage application.
  Newborn Stress Scale: The newborn stress scale developed by Ceylan and Bolışık consists of a total of 24 items in a 3-point Likert type. The scale items include 8 subgroups including facial expression, body color, respiration, activity level, consolability, muscle tone, extremities and posture, and each subgroup is evaluated between 0-2 points in scoring. The minimum score from the scale is zero and the maximum score is 16. As the score increases, the baby's stress level increases.
Salivary Cortisol Level | The newborn baby's salivary cortisol sample will be taken between 05-09 in the morning on the 1st and 4th days of the study.
  The newborn baby's saliva sample will be collected using the Salimetrics SalivaBio Infant's Swab (SIS). To collect a saliva sample, the swab will be held under the tongue and at the corners of the mouth for 60-90 seconds to obtain saliva and placed in the storage tube.
Comfort Score | Every day of the study for 3 days, the newborn's comfort level will be evaluated with the newborn comfort behavior scale 5 minutes before the first massage application and 5 minutes after the third massage application.
  Newborn Comfort Behavior Scale: The newborn comfort behavior scale, whose validity and reliability was established by Kahraman, Başbakkal and Yalaz (2014), is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension and muscle tone. is the scale. Each item in the scale is scored from 1 to 5. It is evaluated based on the total score. The lowest score that can be obtained from the Newborn Comfort Behavior Scale is 6 and the highest score is 30. It is emphasized that if the total score of the scale is between 9-13, the baby is comfortable, if it is between 14-30, the baby is in pain or distress, the baby is uncomfortable and needs interventions to provide comfort.
Bilirubin Level | Every day of the study for 3 days, the newborn baby's bilirubin level will be measured twice a day (before the first massage application and after the third massage application) with a non-invasive bilirubin device
  Non-invasive bilirubin device: Non-invasive bilirubin device is a measuring device that measures babies' serum bilirubin non-invasively through the skin and has a measurement range of at least 0.0-20mg/dL. Bilirubin levels of newborns will be measured with this tool and recorded in the Monitoring Form.
Nutrient ıntake amount | It will be monitored every day of the study for 3 days.
  Nutrient ıntake amount will be monitored on the daily nurse observation form.
Abdominal Circumference Measurement | Every day of the study for 3 days, abdominal circumference will be measured with the same tape measure.
  Abdominal circumference will be measured with the same tape measure immediately before and after each massage application during the research.
Defecation Frequency | It will be monitored every day of the study for 3 days.
  Defecation frequency will be monitored on the daily nurse observation form.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Bayat, Study Director — TC Erciyes Universty

IPD SHARING:
Plan to Share IPD: No